CLINICAL TRIAL: NCT07366346
Title: Effectiveness of a Brief Compensatory Cognitive Training Protocol in People With Mild Cognitive Impairment
Brief Title: Brief Cognitive Training for Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202501616
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: MCI; Mild Cognitive Impairment; Mild Cognitive Impairment (MCI)
Keywords: cognitive training; compensatory cognitive training; mild cognitive impairment; cognitive decline; cognitive intervention; cognitive strategies; group intervention; everyday functioning; cognition; brain health; dementia prevention; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief cognitive training (5 weeks) (Experimental): Participants in this group will attend the brief, five-week version of cognitive training
  Interventions: Behavioral: Brief Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (bME-CCT-MCI)
- Full cognitive training (8 weeks) (Active Comparator): Participants in this group will attend the full, eight-week version of cognitive training
  Interventions: Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT-MCI)

INTERVENTIONS:
Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT-MCI) — ME-CCT-MCI is a publicly available manual for people with mild cognitive impairment (MCI) which has shown effectiveness in improving cognitive performance. Course material will be from the manualized protocol by Huckans and Twamley et al. (2018). The manual includes brief motivational interviewing techniques and modules designed to support behaviors that enhance cognition, such as physical activity, strategies to support learning and memory, mindfulness, and the use of day planners and calendars. It includes the use of frequent breaks, and at-home practice exercises. Each weekly session will be completed in groups of 8-10 participants, and will be led by trained intervention leaders.
  Arms: Full cognitive training (8 weeks)
Behavioral: Brief Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (bME-CCT-MCI) — bME-CCT-MCI is a shortened version of the full ME-CCT-MCI, from eight weeks to five weeks. It preserves core principles of cognitive compensation and habit learning, with a booster summary session in week 5 to reinforce retention. Other than the condensed material, sessions are the same as those in the full ME-CCT-MCI.
  Arms: Brief cognitive training (5 weeks)

SUMMARY:
The goal of this clinical trial is to develop a five-week cognitive training intervention for people with Mild Cognitive Impairment (MCI). The main question it aims to answer is:

• Is five weeks of training as good as eight weeks in improving cognition, quality of life, daily functioning, and mood, and in reducing caregiver burden? Researchers will compare five weeks of cognitive training to eight weeks of training to see if the shorter version is as effective as the full training.

Participants will: [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

* Complete a virtual screening visit with a study partner (typically a family member, roommate, or close friend) to determine eligibility to participate in the study
* Complete some in-person tests of memory and thinking on the University of Florida's campus, and some questionnaires
* Attend weekly two-hour group cognitive training sessions with a trained group leader on campus, for five or eight weeks
* Redo the in-person questionnaires and tests of memory and thinking immediately after completing the training, and three months after completing the training

DETAILED DESCRIPTION:
Background:

In 2024, Alzheimer's disease and other dementias were estimated to cost approximately $360 billion, and these costs are only expected to grow, with estimates rising over $1 trillion by 2050. Although research in pharmacological and brain stimulation interventions is growing, The purpose of this project is to assess the efficacy of brief and full compensatory cognitive training protocols in people diagnosed with Mild Cognitive Impairment (MCI), a state often thought of as a transitory stage between normal aging and dementia. According to the Alzheimer's Association, one in three older adults dies with Alzheimer's disease or another dementia. Research on dementia interventions is growing, with research on neurotransmitter augmentation showing cognitive improvement, and more recently, brain stimulation showing gains in memory and general cognition. However, brain stimulation is not yet approved by the U.S. Food and Drug Administration, and eligibility for anti-amyloid medications is restricted to patient with Alzheimer's Disease pathology and low risk profiles, severely limiting accessibility for many patients. Cognitive rehabilitation is a low-cost solution that is not restricted to patients meeting certain requirements or with a specific etiology and can be utilized by any trained clinician. Cognitive training and rehabilitation is typically categorized as either restorative or compensatory. Restorative training involves repetitive tasks targeting specific cognitive domains (e.g., attention, memory) by harnessing the brain's plasticity and is often completed via computer-based exercises, but often lacks generalizability. Compensatory rehabilitation focuses on individualized strategies that use alternative cognitive processes and supportive aids to compensate for impairment rather than improving it. Cognitive training generally improves quality of life more than pharmacological treatments, and cognitive rehabilitation is particularly effective at improving functional ability and reducing caregiver burden.

Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) is a compensatory cognitive training program which uses cognitive strategies to improve cognition and daily functioning. Originally developed for veterans with traumatic brain injury, it includes a publicly available manual for people with MCI called Motivationally Enhanced Compensatory Cognitive Training for MCI (ME-CCT-MCI), which has shown effectiveness in improving cognitive performance. This program consists of eight two-hour sessions delivered once per week over eight weeks. However, approximately 74% of providers report modifying CogSMART by combining, modifying, or omitting exercises. Despite this, no research to date has examined the effectiveness of an abbreviated version, though evidence from shorter-term psychotherapy suggests it is not significantly less effective than longer-term approaches. This study will develop and implement a five-session version of ME-CCT-MCI, to reduce time burdens and increase accessibility, feasibility, and adherence for patients, caregivers, and providers.

This proposal advances current science in several ways. First, it further validates the ME-CCT-MCI manual. Though extensive research supported the development of this manual, there have only been a small number of studies that have since validated its use. Of these studies, two cite the Indian Adapted ME-CCT-MCI, two study telehealth adaptations, and the last focuses on physical activity and sleep, with no evaluation of its effect on cognition. Second, creating and testing a brief version of this manual allows for improved accessibility. Third, the use of an extensive neuropsychological battery (the National Alzheimer's Coordinating Center Uniform Data Set [NACC-UDS]) allows assessment of improvement in specific cognitive domains. Though research has shown that compensatory cognitive rehabilitation is beneficial to cognition, there is less clear evidence of the specific pattern of effect on cognitive domains, which may help inform clinical decision making in determining which patients may benefit the most from this intervention. Fourth, this study will investigate what participant factors (i.e., education, baseline cognition, and hippocampal volume) predict benefit of intervention, further determining which patients may benefit from this intervention and contributing to future development of personalized medicine.

Specific Aims:

Aim 1: Determine the impact of a feasibility-focused five-session version compared to the full version of the ME-CCT-MCI on cognition, quality of life, daily functioning, mood, and caregiver burden. H1.1: The brief version will not have a worse benefit to participants than the full version of ME-CCT-MCI. H1.2: Benefits of intervention in both groups will be seen particularly in quality of life, activities of daily living, and caregiver burden. Within cognitive domains, there will be particular benefit to learning and executive functioning compared to processing speed and language.

Aim 2 (Exploratory): Investigate individual characteristics that predict cognitive benefits of intervention. Assess moderation effects of demographic factors, baseline cognitive scores, and neuroimaging (Magnetic Resonance Imaging [MRI]) on predicting a greater benefit of intervention on cognition. H2.1: Participants with lower education levels and poorer baseline cognition will show less cognitive benefit from the interventions compared to those with higher education and better baseline performance. H2.2: Lower hippocampal volume will similarly be associated with reduced benefit to cognition compared to those with greater hippocampal volume.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 65 years of age
* Have the ability to speak and understand English
* Time and willingness to commit to the completion of this study
* Availability of a study partner (typically a relative, spouse, offspring, or roommate) for initial and post-intervention testing
* Evidence of a previous MCI diagnosis from participation in another Center for Cognitive Aging and Memory (CAM) study, or a global Clinical Dementia Rating scale (CDR) score of 0.5 and cognitive performance of <26 on the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality) or any history of agitation and/or delirium
* Hearing or vision deficits that would interfere with standardized cognitive assessment or participation in study interventions: i.e. inability to hear through headphones (with or without hearing aids), macular degeneration or other significant diseases that cause severe loss of vision. If vision is corrected with lenses to appropriate levels, then participant will be eligible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in cognition | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the National Alzheimer's Coordinating Center Uniform Data Set version 4 (NACC-UDSv4). This full neuropsychological assessment consists of neuropsychological tests including: Montreal Cognitive Assessment (MoCA), Craft Story 21, Benson Complex Figure, Number Span Test (Forward and Backward), Category Fluency, Trail Making Test, Verbal Fluency: Phonemic Test, Rey Auditory Verbal Learning Test (RAVLT), and Multilingual Naming Test (MINT). On most of these tasks a higher score indicates better cognition, except for on Trail Making Test, where a lower score indicates faster time (better cognition).
Change in quality of life | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Quality of Life in Alzheimer's Disease (QOL-AD), completed by participant and study partner, where higher scores indicate better quality of life (range 13-52).
Change in subjective cognition | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 Cognitive Function 8a, a self-report cognitive functioning questionnaire, where a higher score indicates better reported cognition (range 8-40).
Change in daily functioning | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the National Alzheimer's Coordinating Center (NACC) Functional Assessment Scale (FAS), completed by the study partner, where a lower score indicates more independence (range 0 to 30).
Change in anxiety | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Generalized Anxiety Disorder 7-item (GAD-7) scale, a self-report questionnaire of anxiety, where higher scores indicate higher levels of anxiety (range 0 to 21).
Change in depression | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Geriatric Depression Scale (GDS), a self-report questionnaire of depression, where higher scores indicate higher levels of depression (range 0 to 15).
Change in caregiver burden | Baseline, end of treatment (5 or 8 weeks after baseline, up to 7 or 10 weeks after baseline), and three months after end of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Zarit Burden Interview (ZBI), completed by study partner, where a higher score indicates higher burden (range 0 to 48).

SECONDARY OUTCOMES:
Individual characteristics that predict cognitive benefits of intervention | Baseline
  Assess moderation effects of education, baseline cognitive scores, and neuroimaging (Magnetic Resonance Imaging [MRI]) on predicting a greater benefit of intervention on cognition.

OTHER OUTCOMES:
Treatment satisfaction | End of treatment (18 or 21 weeks after baseline, up to 20 or 23 weeks after baseline)
  As assessed by the Client Satisfaction Questionnaire (CSQ-8), completed by participant and study partner, where a higher score indicates greater satisfaction (range 8 to 32).

CONTACTS AND LOCATIONS:
Overall Officials: Cameron K Perrin, M.S., Principal Investigator — University of Florida; Joseph M Gullett, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The cognitive assessment data will be deidentified and made publicly available upon study completion. Permission to disseminate the neuroimaging data to a larger audience has not been granted so this will not be included in the publicly available dataset.
  A data dictionary will be available accompanying the cognitive assessment data. The manual for the compensatory training intervention (Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment) is already publicly available, and any changes made in this study to create a brief version will also be shared.
  Code created to analyze the results data (in R, python, or MATLAB) will be cleaned for comprehension and shared to support replication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made fully accessible after the study is completed and published, and before the PI (Cameron Perrin) has graduated in 2028. Open Science Framework is designed to support long-term preservation of research data, so the data will be accessible for as long as this service is available.
Access Criteria: Access to this scientific data will not be controlled and will be made publicly available on Open Science Framework.

REFERENCES:
- [Background] Huckans M, Hutson L, Twamley E, Jak A, Kaye J, Storzbach D. Efficacy of cognitive rehabilitation therapies for mild cognitive impairment (MCI) in older adults: working toward a theoretical model and evidence-based interventions. Neuropsychol Rev. 2013 Mar;23(1):63-80. doi: 10.1007/s11065-013-9230-9. Epub 2013 Mar 8. PMID 23471631
- [Background] Lindamer L, Almklov E, Pittman JOE, Shi S, Maye J, Jak A, Twamley E, Rabin B. Multi-method study of the implementation of Cognitive Symptom Management and Rehabilitation Training (CogSMART) in real-world settings. BMC Health Serv Res. 2022 Dec 17;22(1):1542. doi: 10.1186/s12913-022-08941-z. PMID 36528588
- [Background] Juul S, Jakobsen JC, Jorgensen CK, Poulsen S, Sorensen P, Simonsen S. The difference between shorter- versus longer-term psychotherapy for adult mental health disorders: a systematic review with meta-analysis. BMC Psychiatry. 2023 Jun 16;23(1):438. doi: 10.1186/s12888-023-04895-6. PMID 37328755
- [Background] Stypulkowski K, Anquillare E, Twamley EW, Thayer RE. Feasibility of a Telehealth Compensatory Cognitive Training Program for Older Adults with Mild Cognitive Impairment. Clin Gerontol. 2024 Jan-Dec;47(1):17-25. doi: 10.1080/07317115.2023.2213694. Epub 2023 May 17. PMID 37195804
- [Background] Beekly DL, Ramos EM, Lee WW, Deitrich WD, Jacka ME, Wu J, Hubbard JL, Koepsell TD, Morris JC, Kukull WA; NIA Alzheimer's Disease Centers. The National Alzheimer's Coordinating Center (NACC) database: the Uniform Data Set. Alzheimer Dis Assoc Disord. 2007 Jul-Sep;21(3):249-58. doi: 10.1097/WAD.0b013e318142774e. PMID 17804958
- [Background] Huang HC, Tseng YM, Chen YC, Chen PY, Chiu HY. Diagnostic accuracy of the Clinical Dementia Rating Scale for detecting mild cognitive impairment and dementia: A bivariate meta-analysis. Int J Geriatr Psychiatry. 2021 Feb;36(2):239-251. doi: 10.1002/gps.5436. Epub 2020 Oct 9. PMID 32955146
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Lai JS, Wagner LI, Jacobsen PB, Cella D. Self-reported cognitive concerns and abilities: two sides of one coin? Psychooncology. 2014 Oct;23(10):1133-41. doi: 10.1002/pon.3522. Epub 2014 Apr 3. PMID 24700645
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Gullett JM, Albizu A, Fang R, Loewenstein DA, Duara R, Rosselli M, Armstrong MJ, Rundek T, Hausman HK, Dekosky ST, Woods AJ, Cohen RA. Baseline Neuroimaging Predicts Decline to Dementia From Amnestic Mild Cognitive Impairment. Front Aging Neurosci. 2021 Dec 7;13:758298. doi: 10.3389/fnagi.2021.758298. eCollection 2021. PMID 34950021
- [Background] Twamley EW, Jak AJ, Delis DC, Bondi MW, Lohr JB. Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) for veterans with traumatic brain injury: pilot randomized controlled trial. J Rehabil Res Dev. 2014;51(1):59-70. doi: 10.1682/JRRD.2013.01.0020. PMID 24805894
- [Background] Paggetti A, Druda Y, Sciancalepore F, Della Gatta F, Ancidoni A, Locuratolo N, Piscopo P, Vignatelli L, Sagliocca L, Guaita A, Secreto P, Stracciari A, Caffarra P, Vanacore N, Fabrizi E, Lacorte E; Italian Dementia Guideline Working Group. The efficacy of cognitive stimulation, cognitive training, and cognitive rehabilitation for people living with dementia: a systematic review and meta-analysis. Geroscience. 2025 Feb;47(1):409-444. doi: 10.1007/s11357-024-01400-z. Epub 2024 Nov 1. PMID 39485657
- [Background] Luxton D, Thorpe N, Crane E, Warne M, Cornwall O, El-Dalil D, Matthews J, Rajkumar AP. Systematic review of the efficacy of pharmacological and non-pharmacological interventions for improving quality of life of people with dementia. Br J Psychiatry. 2026 Jan;228(1):55-67. doi: 10.1192/bjp.2025.11. Epub 2025 Apr 1. PMID 40166965
- [Background] Gopi Y, Wilding E, Madan CR. Memory rehabilitation: restorative, specific knowledge acquisition, compensatory, and holistic approaches. Cogn Process. 2022 Nov;23(4):537-557. doi: 10.1007/s10339-022-01099-w. Epub 2022 Jul 5. PMID 35790619
- [Background] Jak A. Cognitive Rehabilitation for Adults with a History of Traumatic Brain Injury. Neurol Clin. 2024 Nov;42(4):931-941. doi: 10.1016/j.ncl.2024.05.015. Epub 2024 Jun 15. PMID 39343485
- [Background] Fox NC, Belder C, Ballard C, Kales HC, Mummery C, Caramelli P, Ciccarelli O, Frederiksen KS, Gomez-Isla T, Ismail Z, Paquet C, Petersen RC, Perneczky R, Robinson L, Sayin O, Frisoni GB. Treatment for Alzheimer's disease. Lancet. 2025 Sep 27;406(10510):1408-1423. doi: 10.1016/S0140-6736(25)01329-7. Epub 2025 Sep 22. PMID 40997839
- [Background] Majdi A, van Boekholdt L, Sadigh-Eteghad S, Mc Laughlin M. A systematic review and meta-analysis of transcranial direct-current stimulation effects on cognitive function in patients with Alzheimer's disease. Mol Psychiatry. 2022 Apr;27(4):2000-2009. doi: 10.1038/s41380-022-01444-7. Epub 2022 Feb 3. PMID 35115703
- [Background] Heidebrink JL, Paulson HL. Lessons Learned from Approval of Aducanumab for Alzheimer's Disease. Annu Rev Med. 2024 Jan 29;75:99-111. doi: 10.1146/annurev-med-051022-043645. PMID 38285515
- [Background] Olivares D, Deshpande VK, Shi Y, Lahiri DK, Greig NH, Rogers JT, Huang X. N-methyl D-aspartate (NMDA) receptor antagonists and memantine treatment for Alzheimer's disease, vascular dementia and Parkinson's disease. Curr Alzheimer Res. 2012 Jul;9(6):746-58. doi: 10.2174/156720512801322564. PMID 21875407
- [Background] Danysz W, Parsons CG. The NMDA receptor antagonist memantine as a symptomatological and neuroprotective treatment for Alzheimer's disease: preclinical evidence. Int J Geriatr Psychiatry. 2003 Sep;18(Suppl 1):S23-32. doi: 10.1002/gps.938. PMID 12973747
- [Background] Anand P, Singh B. A review on cholinesterase inhibitors for Alzheimer's disease. Arch Pharm Res. 2013 Apr;36(4):375-99. doi: 10.1007/s12272-013-0036-3. Epub 2013 Feb 24. PMID 23435942
- [Background] Birks J. Cholinesterase inhibitors for Alzheimer's disease. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD005593. doi: 10.1002/14651858.CD005593. PMID 16437532
- See also: Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT-MCI) manual — https://cogtale.org/wp-content/uploads/2023/05/Motivationally-Enhanced-Compensatory-Cognitive-Training-for-MCI-2.pdf